CLINICAL TRIAL: NCT00386737
Title: Development of a Breath Analyzer for Asthma Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ekips Technologies (Industry)
Collaborators: American Lung Association (Other)
Other Study IDs: NIH-2-R44-HL070344-02
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2006-10

CONDITIONS: Asthma
Keywords: Asthma; Breath Testing; Laser Spectroscopy; eNO; Nitric Oxide; Lower Airway Inflammation; Carbon Dioxide; CO2
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Annually, asthma is responsible for 1 million emergency room visits, 400,000 hospitalizations, and 5000 deaths according to the NHLBI. In addition, 10 million missed school-days per year and 100 million days of restricted activity are attributed to this disease. While there is no known cause or cure for asthma, recent studies have shown that hospitalizations and emergency room visits can be reduced by as much as 78% and 73%, respectively, when the disease is properly managed. According to the EPA, the occurance of children with asthma more than doubled the rate of two decades ago; in 2001 the percentage of asthmatic children was 8.7% (6.3 million children).

Properly managing asthma is nontrivial and can often require an asthma specialist. The difficulty in diagnosing and managing asthma lies primarily in the lack of available clinical technologies capable of assessing airway inflammation, an early and persistent component of asthma. Accordingly, the National Institutes of Health (NIH) guidelines for the diagnosis and management of asthma strongly recommend long term anti-inflammatory therapies, such as oral or inhaled corticosteroids, to reverse airway inflammation in an effort to prevent irreversible airway damage, termed "airway remodeling". The medical community has expressed the need for more objective and noninvasive measures of airway inflammation for diagnosing asthma and monitoring the effectiveness and compliance of anti-inflammatory therapies.

The clinical research plan is designed to evaluate airway inflammation associated with asthma. In this human subjects study, a non-invasive exhaled breath analysis sensor, called the Breathmeter, will be used to measure eNO concentrations in children and adults (ages 4-65) with a broad range of respiratory disorders as well as those with no known respiratory disorders. Breath donations will be simple and straightforward presenting little to no discomfort to volunteers.

DETAILED DESCRIPTION:
The study plan is divided into two sections: in-clinic studies and large-scale outreach screening.

(A). Clinical Studies The clinical study is intended to obtain data characterizing eNO concentrations within individual groups of subjects listed in the inclusion criteria. The type of this study is "non-invasive", and the study design is "diagnosis/ treatment monitoring, and efficacy". The study will seek to recruit subjects who fall into one of the categories listed in the inclusion criteria below. The number of subjects (n) to be recruited for each category is given and is estimated based on the past number of subjects mainly at the Ekips Technologies, The Oklahoma Allergy & Asthma Clinic, and the Norman Lung Center sites.

Inclusion Criteria (Total Number of Subjects, n = 700)

Both genders are eligible for this study:

1. Healthy subjects (n=120)
2. Asthma (Total n=450) [diagnosed according to NHLBI/ NAEPP Guidelines (1998)]

   1. Non-treated or B2-agonist treated asthmatics (n=150),
   2. Glucocorticoid treated asthmatics, (n=150),
   3. Leukotriene Antagonist treated asthmatics, (n=75),
   4. Glucocorticoid and Leukotriene Antagonists treated asthmatics, (n= 75).
3. Acute respiratory illnesses (n=65

   a) Sinusitis (Acute and Chronic), b) Influenza, c) Common cold, d)Pneumonia, e)Related symptoms, but no diagnosis.
4. Allergies (n=65) a) Atopic dermatitis, b) Allergic rhinitis, c) Seasonal allergies.

Healthy Subjects Recruiting

Healthy subjects will be recruited from visitors and patients at the study sites. Visitors may include relatives or friends accompanying patients. Healthy employees at the study sites may be asked to participate in the study. Patients, visitors, and employees will be told that do not have to participate if they do not want to.

Exclusion Criteria

Subjects younger than 4 and older than 65 will be excluded from the study. Pregnant women will also be excluded from the study.

Duration of Participation

For each visit, the participant in the study will be asked to donate up to 3 breath samples for the first visit. The total time required for breath donations and measurements will be about 5 minutes. An additional five minutes of a subject's time are needed to complete a short interview if the information needed is not already available.

Asthmatic or suspected asthmatic patients, both treated and non-treated will be asked to donate breath during additional visits if convenient. Follow-up measurements may be performed during regularly scheduled office visits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (n=120)
* Asthma (Total n=450) [diagnosed according to NHLBI/ NAEPP Guidelines (1998)]

  * Non-treated or B2-agonist treated asthmatics (n=150),
  * Glucocorticoid treated asthmatics, (n=150),
  * Leukotriene Antagonist treated asthmatics, (n=75),
  * Glucocorticoid and Leukotriene Antagonists treated asthmatics, (n= 75).
* Acute respiratory illnesses (n=65

  * Sinusitis (Acute and Chronic),
  * Influenza,
  * Common cold,
  * Pneumonia,
  * Related symptoms, but no diagnosis.
* Allergies (n=65)

  * Atopic dermatitis,
  * Allergic rhinitis,
  * Seasonal allergies.

Exclusion Criteria:

* Younger than 4
* Older than 65
* Pregnant

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000
Dates: Start 2004-09; Study Completion 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: Khosrow Namjou, Ph.D., Principal Investigator — Ekips Technologies, Inc.
Locations (1):
- Ekips Technologies, Inc., Norman, Oklahoma, United States